CLINICAL TRIAL: NCT05714137
Title: Evaluation of the Effect of Proximal Massage and Fist Clenching in Reducing the Risk of Phlebitis From Peripheral Venous Catheter
Brief Title: Reducing the Risk of Phlebitis From Peripheral Venous Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, SERAP GÜNGÖR, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4819
Record Dates: First submitted 2023-01-08; First posted 2023-02-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Phlebitis
Keywords: Phlebitis; Peripheric venous catheter; Nursıng Care; Palm fisting; Proximal massage
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Intervention Model Description: two groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proximal massage and fist clenching (Experimental): The experimental group of 36 patients underwent proximal massage and fist clenching after IV insertion. Proximal massage: For a total of 5 to 10 minutes, twice daily for 4 days, between 30 seconds- 1 minute in sessions of approximately 20 strokes, a light massage is administered utilizing the palm surfaces of the fingers. Fist Clenching : Under the researcher's supervision, participants in the activity known as palm fisting squeeze a soft palm ball 20 times in each of twice a day for four days, lasting between 30 seconds - 1 minute. The Peripheral Venous Catheter-Related Phlebitis Risk Scale, the Phlebitis Diagnostic Scale, and the Patient Information Form were employed right after following PVC (0. hour). The Phlebitis Diagnostic Scale was used for 96 hours to assess the patient's vascular access at the 24th, 48th, 72nd, and 96th hours.
  Interventions: Behavioral: Evaluation of the Effect of Proximal Massage and Fist Clenching in Reducing the Risk of Phlebitis From Peripheral Venous Catheter
- Standard care for PVC (No Intervention): The standard care group of 36 patients received typical nursing PVC care. Standard nurse PVC care: Only standard PVC care and follow-up were provided. It was carefully avoided that the patients would interact with one another or be in the same patient room. The Peripheral Venous Catheter-Related Phlebitis Risk Scale, the Phlebitis Diagnostic Scale, and the Patient Information Form were employed right after following PVC (0. hour). The Phlebitis Diagnostic Scale was used for 96 hours to assess the patient's vascular access at the 24th, 48th, 72nd, and 96th hours.

INTERVENTIONS:
Behavioral: Evaluation of the Effect of Proximal Massage and Fist Clenching in Reducing the Risk of Phlebitis From Peripheral Venous Catheter — Proximal massage: For a total of 5 to 10 minutes, twice daily for 4 days, between 30 seconds- 1 minute in sessions of approximately 20 strokes, a light massage is administered utilizing the palm surfaces of the fingers.
  Fist Clenching : Under the researcher's supervision, participants in the activity known as palm fisting squeeze a soft palm ball 20 times in each of 2 days a day for four days, lasting between 30 seconds - 1 minute.
  Arms: Proximal massage and fist clenching

SUMMARY:
Nurses frequently use peripheral venous catheters in hospitals to provide medications and fluids for therapeutic and diagnostic purposes. Peripheral venous catheter use brought various problems, including phlebitis, infiltration, extravasation, ecchymosis, thrombophlebitis, and embolism, in addition to being a regularly utilized nursing practice. The literature used techniques like heat application, fist clenching, and proximal massage to lower the risk of thrombophlebitis and associated problems.

DETAILED DESCRIPTION:
Between October and November 2022, individuals who received orthopedic care at a state hospital and had peripheral venous catheters participated in the trial as a randomized controlled experimental study. The control group received routine nursing care, while the experimental group received proximal massage and palm fist exercises. The numbers used to identify the control and experimental groups were drawn at random from a table of random numbers, and each group had 36 patients. The researcher used the "Patient Information Form," "Plebitis Risk Scale Due to Peripheral Venous Catheter," and "Plebitis Diagnostic Scale" to collect data using in-person interviews and observational methods. The p value for statistical significance is p<0.05. Proximal massage: For a total of 5 to 10 minutes, twice daily for 4 days, between 30 seconds- 1 minute in sessions of approximately 20 strokes, a light massage is administered utilizing the palm surfaces of the fingers. Under the researcher's supervision, participants in the activity known as fist clenching squeeze a soft palm ball 20 times in each of twice a day for four days, lasting between 30 Seconds - 1 minute.

ELIGIBILITY:
Inclusion Criteria:

* Patients who volunteered to participate in the study,
* Who are over 18 years old,
* Having no barriers to written and verbal communication in Turkish,
* IV treatment was applied during the hospitalization period and IV treatment was recently started,
* Patients with IV cannula in the upper extremity
* In the last six months before hospitalization, IV treatment was not applied,
* A maximum of 2 IV attempts should be made on a patient.
* Patients without chronic dermatological and/or vascular disease.

Exclusion Criteria:

* Patients who did not volunteer to participate in the study, unconscious patients,
* IV attempts were made to the same patient more than 4 times in total,
* Patients with IV cannula in the lower extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Phlebitis Assessment Scale | Within 96 hours, the development of PVC-related phlebitis will be evaluated.
  The scale has five ratings as follows. Phlebitis with this scale: Grade 0: no symptoms, Grade 1: redness and/or pain at the catheter insertion site, Grade 2: redness, pain and/or edema at the catheter insertion site, Grade 3: redness, pain and/or edema at the catheter insertion site , red line, cable-like palpation of the vein, Grade 4: redness, pain and/or edema at the catheter insertion site, red line, cable-like palpation of the vein and if it is longer than 2.5 cm, it is considered as purulent discharge.

SECONDARY OUTCOMES:
Peripheral Venous Catheter-Related Phlebitis Risk Scale | Within the first 24 hours, the patient will be assessed using the Peripheral Venous Catheter-Associated Phlebitis Risk Scale.
  The scale consists of 14 items and three sub-dimensions. There are 3 items in the Individual Risk Factors sub-dimension, 6 items in the Chemical Risk Factors sub-dimension, and 5 items in the Mechanical Risk Factors sub-dimension. The scale has a 2-point rating and is designed to calculate the score for each item as "Yes=2 points" and "No=1 points". There is no reverse item in the scale. An increase in the score obtained from the scale indicates that the risk of phlebitis due to peripheral venous catheters increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam University, Karaman, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heng SY, Yap RT, Tie J, McGrouther DA. Peripheral Vein Thrombophlebitis in the Upper Extremity: A Systematic Review of a Frequent and Important Problem. Am J Med. 2020 Apr;133(4):473-484.e3. doi: 10.1016/j.amjmed.2019.08.054. Epub 2019 Oct 10. PMID 31606488
- [Background] Lv L, Zhang J. The incidence and risk of infusion phlebitis with peripheral intravenous catheters: A meta-analysis. J Vasc Access. 2020 May;21(3):342-349. doi: 10.1177/1129729819877323. Epub 2019 Sep 23. PMID 31547791
- [Background] Zingg W, Pittet D. Peripheral venous catheters: an under-evaluated problem. Int J Antimicrob Agents. 2009;34 Suppl 4:S38-42. doi: 10.1016/S0924-8579(09)70565-5. PMID 19931816
- [Derived] Tosun B, Gungor S, Agkale E, Andi S. Evaluation of the effect of proximal massage and palm fisting in reducing the risk of peripheral venous catheter-related phlebitis: randomized control study. Eur J Cardiovasc Nurs. 2024 Sep 5;23(6):644-651. doi: 10.1093/eurjcn/zvae024. PMID 38366675